CLINICAL TRIAL: NCT01130142
Title: A Phase 1b/2 Study Evaluating IPI-926 in Combination With Gemcitabine in Patients With Metastatic Pancreatic Cancer
Brief Title: A Study Evaluating IPI-926 in Combination With Gemcitabine in Patients With Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Infinity Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IPI-926-03
Record Dates: First submitted 2010-04-21; First posted 2010-05-25 (Estimated); Last update posted 2017-03-06 (Actual); Status verified 2017-03

CONDITIONS: Metastatic Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — IPI-926; Gemcitabine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Phase 2) (Active Comparator): IPI-926 in combination with gemcitabine
  Interventions: Drug: IPI-926 plus gemcitabine
- Arm 2 (Phase 2) (Placebo Comparator): Placebo in combination with gemcitabine
  Interventions: Drug: IPI-926 plus gemcitabine; Drug: Placebo plus gemcitabine

INTERVENTIONS:
Drug: IPI-926 plus gemcitabine — Daily IPI-926 (oral) at 160 mg plus gemcitabine (infusion) at 1000 mg/m2 once weekly for 3 weeks of a 28 day cycle
  Other Names: IPI-926; Hedgehog pathway inhibitor; Hedgehog
Drug: Placebo plus gemcitabine — Daily Oral placebo/IPI-926 160 mg plus gemcitabine infusion at 1000 mg/m2 once every 3 weeks in a 28 day cycle
  Other Names: Gemcitabine; Hedgehog; Hedgehog pathway inhibitor; Gemzar
  Arms: Arm 2 (Phase 2)

SUMMARY:
Study IPI-926-03 is a Phase 1b/2 clinical trial to evaluate IPI 926 in combination with gemcitabine in patients with previously untreated metastatic pancreatic cancer. Phase 1b is designed as a dose escalation study. Once the maximum tolerated dose of IPI-926 in combination with gemcitabine is established in the Phase 1b portion of the study, the Phase 2 portion will commence.

Phase 2 is designed as a randomized, double-blind (investigator/patient), placebo-controlled study. There is no cross-over option for patients in either arm of the Phase 2 (i.e., there is no option for patients receiving placebo to cross-over to IPI-926).

DETAILED DESCRIPTION:
IPI 926 is an inhibitor of the Hedgehog Pathway. IPI-926 in combination with gemcitabine may improve therapeutic outcomes in patients with pancreatic cancer. Infinity is conducting a Phase 1b/2 clinical trial to evaluate the safety and efficacy of IPI-926 in combination with gemcitabine in patients with previously untreated metastatic pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age
* Pathologically confirmed metastatic pancreatic adenocarcinoma
* At least 1 radiologically evaluable metastatic lesion (RECIST 1.1).
* ECOG 0 or 1
* Life expectancy ≥3 months.
* All women of child bearing potential, all sexually active male patients, and partners of patients must agree to use adequate methods of birth control
* Ability to adhere to the study visit schedule
* Voluntarily signed an informed consent form

Exclusion Criteria:

* Islet cell, acinar cell carcinoma, non-adenocarcinoma, (i.e., lymphoma, sarcoma), adenocarcinoma originated from biliary tree or cystadenocarcinoma
* Prior treatment with chemotherapy for pancreatic cancer.
* Known central nervous system metastases
* Inadequate hematologic function
* Inadequate hepatic function
* Inadequate renal function
* External (percutaneous) biliary drain
* History of stroke, unstable angina, myocardial infarction, or ventricular arrhythmia requiring medication or mechanical control within the last 6 months.
* Venous thromboembolic event (e.g., pulmonary embolism or deep vein thrombosis) requiring anticoagulation not appropriately anticoagulated or have NCI CTCAE Grade 2 or greater bleeding episode in the 3 weeks prior to administration of IPI-926
* Concurrent administration of the medications or foods known to inhibit CYP3A activity to a clinically relevant degree
* Presence of active infection or systemic use of antibiotics within 72 hours of treatment
* Significant co-morbid condition or disease which in the judgment of the Investigator would place the patient at undue risk or interfere with the study.
* Known human immunodeficiency virus (HIV) positivity
* Known hypersensitivity to gemcitabine, IPI-926, or their excipients
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2010-04; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Evaluation of safety profile including MTD | Once per week for 3 weeks of a 4 week cycle
  To determine the safety profile, including maximum tolerated dose, of IPI-926 plus gemcitabine in patients with previously untreated metastatic pancreatic cancer.
Overall survival comparison | An average of 6 months
  * To compare the overall survival (OS) of patients with previously untreated metastatic pancreatic cancer treated with IPI-926 plus gemcitabine or placebo plus gemcitabine.
  * To evaluate the safety of IPI-926 plus gemcitabine or placebo plus gemcitabine.

SECONDARY OUTCOMES:
Measurement of the maximum plasma concentration (Cmax) and area under the concentration versus time curve (AUC0-t) of IPI-926 and gemcitabine. | During the 3rd week of the first 4 week cycle
  - To evalutate pharmacokinetics (PK) of IPI-926, gemcitabine, and their relevant metabolites.
Comparison of PFS, TTP and ORR | An average of 6 months
  - To compare the progression free survival (PFS), time to progression (TTP) and overall response rate (ORR) of patients treated with IPI-926 plus gemcitabine or placebo plus gemcitabine.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Ross, MD, Study Director — Infinity Pharmaceuticals, Inc.
Locations (28):
- United States (25):
  - Arizona Clinical Research Center, Tucson, Arizona
  - University of California San Diego Medical Center, San Diego, California
  - University of California San Francisco, San Francisco, California
  - Kaiser Permanente, Vallejo, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Kansas City Cancer Center, Overland Park, Kansas
  - Norton Health Care, Louisville, Kentucky
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Columbia University Medical Center, New York, New York
  - Weill Cornell Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - Willamette Valley Cancer Institute and Research Center, Eugene, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Institute of Translational Oncology Research, Greenville, South Carolina
  - Texas Oncology- Bedford, Bedford, Texas
  - Texas Oncology, PA, Dallas, Texas
  - South Texas Oncology and Hematology, San Antonio, Texas
  - Tyler Cancer Center, Tyler, Texas
  - Virginia Oncology Associates, Newport News, Virginia
  - Seattle Cancer Care Alliance, Seattle, Washington
- Canada (3):
  - Cancer Care Manitoba, Winnipeg, Manitoba
  - Toronto Sunnybrook Regional Cancer Centre, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec

REFERENCES:
- [Derived] Kochetkova M, Samuel MS. Differentiation of the tumor microenvironment: are CAFs the Organizer? Trends Cell Biol. 2022 Apr;32(4):285-294. doi: 10.1016/j.tcb.2021.11.008. Epub 2021 Dec 9. PMID 34895986